CLINICAL TRIAL: NCT00557518
Title: A Randomized, Placebo-Controlled Trial of Alagebrium in Patients With Insulin-Dependent Type 1 Diabetes and Microalbuminuria
Brief Title: Study of Alagebrium in Patients With Insulin-Dependent Type 1 Diabetes and Microalbuminuria
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study has been terminated early due to financial constraints.
Sponsor: Synvista Therapeutics, Inc (Industry)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Mark Cooper, Baker Heart Research Institute, Melbourne, Australia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALT-711-0424
Record Dates: First submitted 2007-11-12; First posted 2007-11-14 (Estimated); Last update posted 2009-01-30 (Estimated); Status verified 2009-01

CONDITIONS: Diabetes Mellitus, Type 1; Diabetic Nephropathy
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetic Nephropathies | interventions — alagebrium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Alagebrium
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Alagebrium — 200 mg bid
  Other Names: ALT-711
  Arms: 1
Drug: Placebo — bid
  Arms: 2

SUMMARY:
Based upon the preclinical evidence in models of diabetic nephropathy under conditions approximating both type I and II diabetes, treatment with alagebrium appears to have favorable and advantageous effects on the biochemical, structural, pathological and functional hallmarks of diabetic nephropathy. The renoprotective effects of alagebrium in preclinical models favor the evaluation of this drug in patients with type I diabetes.

DETAILED DESCRIPTION:
This study is a double-blind, randomized, placebo-controlled, parallel design trial enrolling 80 patients (2x40) with Type 1 diabetes and microalbuminuria. Patients will be randomized to either 200 mg Alagebrium twice daily or placebo for a period of 24 weeks after an 8 week run-in period. There will be a 8 week run-out period. All patients will receive ramipril during the entire study period. Efficacy measurements will be performed at baseline, at 12 weeks and at the end of the study. Measurements for albumin:creatinine ratio(mg/g), plasma renin level, collagen markers, AGE related markers and 24 hour blood pressure measurements will also be determined. A total of 9 visits will be performed during the entire study.

ELIGIBILITY:
Inclusion Criteria:

* Insulin-dependent type 1 diabetes
* Age 18-65 years
* Diagnosis of established microalbuminuria
* Blood pressure <140 mm Hg, diastolic blood pressure <90 mm Hg
* HbA1c <10%

Exclusion Criteria:

* Body mass index >40 kg/m2
* Cardiovascular event within 6 months prior to screening
* History of acute myocardial infarction within 12 months prior to screening
* Serum creatinine >1.5 mg/dL
* Receiving chronic nonsteroidal anti-inflammatory therapy
* Receiving antihypertensive therapy except for angiotensin converting enzyme inhibitors or angiotensin receptor blockers
* Any significant systemic illnesses,medical conditions or abnormal laboratory values

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2007-11; Primary Completion 2009-09 (Estimated); Study Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in albumin excretion rate (µg/min) | 24 weeks

SECONDARY OUTCOMES:
Albumin:creatinine ratio(mg/g), plasma renin level, collagen markers, AGE related markers, 24 hour blood pressure determinations | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mark E Cooper, MBBS, PhD, Study Chair — Baker Heart Research Institute, Melbourne, Australia
Locations (6):
- Australia (5):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - International Diabetes Institute, Caulfield, Victoria
  - Dept. of Clinical and Biomedical Science Myers House, Geelong, Victoria
  - Austin Health, Heidelburg, Victoria
  - The Alfred Hospital, Melbourne, Victoria
- Steno Diabetes Center, Gentofte Municipality, Denmark